CLINICAL TRIAL: NCT01790594
Title: Optimization of NULOJIX® (Belatacept) Usage as a Means of Minimizing CNI Exposure in Simultaneous Pancreas and Kidney Transplantation (CTOT-15)
Brief Title: Optimization of NULOJIX® Usage Towards Minimizing CNI Exposure in Simultaneous Pancreas and Kidney Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual within enrollment time period: projected accrual goal not achieved.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network); Rho Federal Systems Division, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-15; U01AI084150 (NIH); NIAID CRMS ID#: 20117 (Other: DAIT NIAID); SDY1433 (Other: ImmPort)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Simultaneous Kidney and Pancreas Transplantation
Keywords: transplantation; kidney; pancreas; immunosuppression; calcineurin inhibitor (CNI)
MeSH Terms: interventions — Abatacept; Methylprednisolone; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunosuppression without Belatacept (Active Comparator): * Induction: 5 day course of methylprednisolone or equivalent;
  * Induction: Anti-thymocyte Globulin (Rabbit);
  * Maintenance Immunosuppression: Tacrolimus (or generic). The site investigator will identify a starting tacrolimus dose at his or her discretion, in order to achieve the target trough levels, no later than 5 days post-transplantation. Tacrolimus dosing will be initiated on the day of surgery or post-operative day 1 depending upon when during the day the surgery is completed, then adjusted to target trough levels of 8-12 ng/ml during the first 24 weeks post-transplant, then adjusted to target trough levels of 5-8 ng/ml thereafter.
  * Maintenance Immunosuppression: Mycophenolate mofetil (or Myfortic (mycophenolate sodium), or generic).
  Interventions: Drug: methylprednisolone; Biological: Anti-thymocyte Globulin (Rabbit); Drug: Tacrolimus; Drug: Mycophenolate mofetil
- Immunosuppression Including Belatacept (Experimental): * Induction: 5 day course of methylprednisolone or equivalent;
  * Induction: Anti-thymocyte Globulin (Rabbit);
  * Maintenance Immunosuppression: Belatacept
  * Maintenance Immunosuppression: Tacrolimus (or generic)- The site investigator will identify a starting tacrolimus dose at his or her discretion, in order to achieve the target trough levels no later than 5 days post-transplantation. Tacrolimus dosing will be initiated on the day of surgery or post-operative day 1 depending upon when during the day the surgery is completed. The dosage will be adjusted to achieve the following therapeutic trough levels: 5-8 ng/ml during the first 24 weeks post-transplant and then 3-5 ng/ml until day 280 (week 40). Subjects may be withdrawn if they meet all the criteria defined below.
  * Maintenance Immunosuppression: Mycophenolate mofetil (or Myfortic (mycophenolate sodium), or generic).
  Interventions: Biological: Belatacept; Drug: methylprednisolone; Biological: Anti-thymocyte Globulin (Rabbit); Drug: Tacrolimus; Drug: Mycophenolate mofetil

INTERVENTIONS:
Biological: Belatacept — The first dose of belatacept will be administered approximately 24-48 hours after the last dose of Anti-Thymocyte Globulin (Rabbit).
  Other Names: NULOJIX
  Arms: Immunosuppression Including Belatacept
Drug: methylprednisolone
  Other Names: Medrol
Biological: Anti-thymocyte Globulin (Rabbit)
  Other Names: Thymoglobulin; ATG (Rabbit)
Drug: Tacrolimus — There may be an opportunity to withdraw tacrolimus at week 40
  Other Names: Prograf
Drug: Mycophenolate mofetil — Mycophenolate mofetil will be administered at a target dose of 1000 mg by mouth twice daily (e.g., BID) beginning on the day of surgery or post-operative day 1 depending upon when during the day the surgery is completed (maximum MMF dosing is 2G per day). MMF will be adjusted based on clinical complications (such as neutropenia). Myfortic® (mycophenolate sodium) may be used as a replacement for MMF. Mycophenolate sodium will be dosed at 720 mg PO BID. Mycophenolate sodium will be adjusted based on clinical complications.
  Other Names: MMF, mycophenolate sodium, CellCept

SUMMARY:
The purpose of this study is to find out if the drug NULOJIX® (belatacept) will minimize the amount of other anti-rejection medications necessary and thereby reduce the long-term side effects caused by the other medications. The researchers also want to learn more about the safety of this treatment and long term health of transplanted pancreases and kidneys.

DETAILED DESCRIPTION:
Transplant recipients have to take anti-rejection medications to prevent their immune systems (the body's natural defense system against illness) from rejecting their new organs. Most patients who receive a transplanted organ must take these anti-rejection medications for the rest of their lives, or for as long as the transplanted organ continues to work. Taking standard anti-rejection medications for a long time can cause serious side effects, including pancreas and kidney damage. There would be a benefit to finding new anti-rejection medications that work just as well, but could lessen the amount of anti-rejection medications that are taken long term.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide written informed consent;
* Candidate for a primary simultaneous kidney and pancreas allograft with random c-peptide <0.3 ng/mL;
* No known contraindications to study therapy using NULOJIX® (belatacept);
* Female subjects of childbearing potential must have a negative pregnancy test upon study entry;
* Female and male participants with reproductive potential must agree to use FDA approved methods of birth control during participation in the study and for 4 months following study completion;
* No donor specific antibodies prior to transplant that are considered to be of clinical significance by the site investigator;
* Negative crossmatch, actual or virtual, or a Panel Reactive Antibodies (PRA) of 0% on historic and admission sera, as determined by each participating study center;
* A documented negative Tuberculosis (TB) test within the 12 months prior to transplant. If documentation is not present at the time of transplantation, and the subject does not have any risk factors for TB, a TB-specific interferon gamma release assay (IGRA) may be performed.

Exclusion Criteria:

* Need for multi-organ transplantation other than a kidney and pancreas;
* Recipient of previous organ transplant;
* Epstein-Barr Virus (EBV) sero-negative recipients or recipients whose EBV serostatus is unknown prior to the time of transplantation;
* Individuals infected by the hepatitis B or C viruses or HIV;
* Individuals who have required treatment with systemic prednisone or other immunosuppressive drugs within 1 year prior to transplant;
* Individuals previously treated with NULOJIX® (belatacept);
* Any condition that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements;
* Use of investigational drugs within 4 weeks of enrollment;
* Known hypersensitivity to mycophenolate mofetil (MMF)or any of the drug's components;
* Administration of live attenuated vaccine(s) within 8 weeks of enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Newell, MD, PhD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco Medical Center, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data is available in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Supporting Information: Study Protocol
Time Frame: On average, data is available within 24 months after database lock for a trial.
Access Criteria: Open access.
  Study's:
  * Accession ID is SDY1433, and
  * Digital Object Identifier (DOI) is : 10.21430/M3CEH2A7ZF
URL: https://www.immport.org/home

REFERENCES:
- [Result] Stock PG, Mannon RB, Armstrong B, Watson N, Ikle D, Robien MA, Morrison Y, Odorico J, Fridell J, Mehta AK, Newell KA. Challenges of calcineurin inhibitor withdrawal following combined pancreas and kidney transplantation: Results of a prospective, randomized clinical trial. Am J Transplant. 2020 Jun;20(6):1668-1678. doi: 10.1111/ajt.15817. Epub 2020 Mar 8. PMID 32039559
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation (CTOT) website — https://www.ctotstudies.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five sites in the United States recruited and enrolled 46 participants into this trial.
Groups:
- Investigational: Induction: Methylprednisolone (MEDROL) was administered at a dose of 500 mg on the day of transplant, and tapered to 250 mg on day 1, 125 mg on day 2, 60 mg on day 3, 30 mg on day 4, and 0 mg on day 5. A target dose of 6 mg/kg over 3 to 4 days of Thymoglobulin was administered via intravenous infusion. Maintenance: Belatacept (NULOJIX) was given at a dose of 10 mg/kg on days 5, 14, 28, 56, and 84. After 84 days participants received 5 mg/kg every 4 weeks until the completion of the trial. Site investigator determined the initial dose of tacrolimus (tac) started on the day of transplant or day 1. Dosing was adjusted to achieve a target trough of 5-8 ng/ml during the first 24 weeks, and adjusted to 3-5 ng/ml until week 40. If eligible, at week 40 tac withdrawal was initiated over a 4-8 week period. Mycophenolate Mofetil (MMF) or equivalent was administered at a target dose of 1000 mg PO or IV BID starting on the day of transplant or day 1.
- Control: Induction: 500 mg of MEDROL was administered on the day of transplant, and tapered to 250 mg on day 1, 125 mg on day 2, 60 mg on day 3, 30 mg on day 4, and 0 mg on day 5. A target dose of 6 mg/kg over 3 to 4 days of Thymoglobulin was administered via intravenous infusion. Maintenance: Site investigator determined the initial dose of tacrolimus (tac) that started on the day of transplant or day 1. Dosing was adjusted to achieve a target trough of 8-12 ng/ml during the first 24 weeks, and adjusted to 5-8 ng/ml thereafter. Mycophenolate Mofetil (MMF) or equivalent was administered at a target dose of 1000 mg PO or IV BID starting on the day of transplant or day 1.
- Enrolled, Not Randomized: Subjects who signed informed consent and were thus enrolled, but were not randomized to study treatment.
Period: Overall Study
Arm/Group | Investigational | Control | Enrolled, Not Randomized
Started | 22 | 21 | 3
Completed | 17 | 18 | 0
Not Completed | 5 | 3 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Transplant was not done | 0 | 0 | 3
Not completed — Terminated prior to week 76 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational | Control | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (7.10) | 38.8 (6.98) | 39.3 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 5 | 8
  White | 18 | 14 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Estimated Glomerular Filtration Rate (eGFR) Calculated for Each Treatment Group Using the CKD-EPI Equation at Wk 52 Post-Transplant
Description: eGFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI):
  * A score of ≥90 means kidney function is normal.
  * A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease.
  * Scores between 30 and 59 indicates moderately reduced kidney function.
  * Scores between 15 and 29 indicate severely reduced kidney function.
  * Scores below 15 indicate very severe or end stage kidney failure.
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population with available data at week 52.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Investigational | Control
Number analyzed (Participants) | 21 | 21
mL/min/1.73m^2 | 77.0 (22.6) | 74.6 (19.7)
Statistical Analysis 1: Comparison: Investigational vs Control; The p-value compares Investigational arm and control arm; Test type: Superiority; p = 0.750, Mixed Models Analysis; Mean Difference (Final Values) = 2.088, 95% CI 2-sided [-11.067 to 15.242]

2. Secondary Outcome: Count of Participants With eGFR < 60 mL/Min/1.73 m^2 Measured by CKD-EPI at Wk 52 Post-Transplant
Description: as for outcome 1
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants | 5 | 5

3. Secondary Outcome: Count of Participants by CKD Stage at Wk 52 Post-Transplant
Description: The stages of Chronic Kidney Disease are defined using the participant's GFR value:
  * Stage 1 if GFR value is ≥90 ( kidney function is normal)
  * Stage 2 if 60 ≤ GFR < 90 (mildly reduced kidney function, pointing to kidney disease)
  * Stage 3A if 45 ≤ GFR < 60*
  * Stage 3B if 30 ≤ GFR < 45*
  * Stage 4 if 15 ≤ GFR < 30 (severely reduced kidney function)
  * Stage 5 if GFR < 15 (severe or end stage kidney failure).
  Stages 3A and 3B indicate moderately reduced kidney function.*
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 21 | 21
Participants
  Stage 1 | 5 | 5
  Stage 2 | 11 | 11
  Stage 3A | 2 | 4
  Stage 3B | 3 | 1
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

4. Secondary Outcome: Count of Participants With Defined CKD Stage 4 or 5 at Wk 52 Post-Transplant
Description: The stages of Chronic Kidney Disease (CKD) are defined using the participant's GFR value:
  * Stage 1 if GFR value is ≥ 90 (kidney function is normal)
  * Stage 2 if 60 ≤ GFR < 90 (mildly reduced kidney function, pointing to kidney disease)
  * Stage 3A if 45 <= GFR < 60*
  * Stage 3B if 30 <= GFR < 45*
  * Stage 4 if 15 ≤ GFR < 30 (severely reduced kidney function)
  * Stage 5 if GFR < 15 (severe or end stage kidney failure).
  Stages 3A abd 3B indicate moderately reduced kidney function.*
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

5. Secondary Outcome: Mean Calculated eGFR Using MDRD 4 Variable Model at Wk 52 Post-Transplant
Description: The estimated Glomerular Filtration Rate (eGFR) was calculated using the Modification of Diet in Renal Disease equation (MDRD):
  * A score of ≥ 90 means kidney function is normal.
  * A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease.
  * Scores between 30 and 59 indicates moderately reduced kidney function.
  * Scores between 15 and 29 indicate severely reduced kidney function.
  * Scores below 15 indicate severe or endstage kidney failure.
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Investigational | Control
Number analyzed (Participants) | 21 | 21
mL/min/1.73m^2 | 68.7 (19.5) | 67.0 (17.6)

6. Secondary Outcome: The Slope of eGFR by CKD-EPI Over Time Based on Serum Creatinine Post-Transplant
Description: The estimated Glomerular Filtration Rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI):
  * A score of ≥ 90 means kidney function is normal.
  * A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease.
  * Scores between 30 and 59 indicates moderately reduced kidney function.
  * Scores between 15 and 29 indicate severely reduced kidney function.
  * Scores below 15 indicate very severe or endstage kidney failure.
  An estimate of the slope, or change over time, in eGFR was produced using standard statistical linear modeling procedures. The estimate was then re-scaled so that it could be interpreted as a change in eGFR per month. Positive numbers indicate increasing kidney function.
  Larger numbers indicate greater change in kidney function.
Time Frame: Day 28 through Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: eGFR change over time (by month)
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
eGFR change over time (by month) | 0.1 (3.1) | -0.1 (2.5)

7. Secondary Outcome: Count of Participants With Successful Discontinuation of Tacrolimus in Recipients Randomized to the Investigational Arm
Description: Participants achieved successful discontinuation if they were able to discontinue (e.g., off tacrolimus therapy completely) over a 4-8 weeks after tacrolimus withdrawal was initiated at week 40.
Time Frame: Week 40 through week 48 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational
Number analyzed (Participants) | 22
Participants | 5

8. Secondary Outcome: Count of Participants With Delayed Graft Function at Wk 52 Post-Transplant
Description: Delayed grafted function is defined as dialysis in the first week on one or more occasions for any indication other than the treatment of acute hyperkalemia in the setting of otherwise acceptable renal function.
Time Frame: Transplant through Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants | 1 | 1

9. Secondary Outcome: Count of Participants With Full Pancreatic Graft Function (Insulin Independent) at Wk 52 Post-Transplant
Description: Participants with full pancreatic graft functions are defined as those that no longer require exogenous insulin therapy.
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 21 | 21
Participants | 19 | 21

10. Secondary Outcome: Count of Participants With Evidence of Partial Pancreatic Graft Function at Week 52 Post-Transplant
Description: C-peptide is a measure of pancreatic function. The definition of partial pancreatic graft function: a fasting C-peptide levels >0.3ng.mL (0.1nmol.L) plus the participant's continued requirement for exogenous insulin or oral hypoglycemic agent(s).
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 18 | 17
Participants | 1 | 0

11. Secondary Outcome: Count of Participants With Evidence of Pancreatic Loss at Week 52 Post-Transplant
Description: C-peptide is a measure of pancreatic function. The definition of pancreatic loss: a C-peptide value of <0.3 ng/mL.
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 18 | 17
Participants | 1 | 0

12. Secondary Outcome: HbA1c at Baseline (Pre-Transplant) Through Wk 52 Post-Transplant
Description: Hemoglobin A1c (HbA1c) measures the average blood glucose levels over 8-12 weeks, thus acting as a useful long-term gauge of blood glucose control:
  * A value below 6.0% reflects normal levels,
  * 6.0% to 6.4% reflects prediabetes, and
  * a value of ≥ 6.5% reflects diabetes.
Time Frame: Baseline (Pre-Transplant) and Days 28, 84, and Weeks 28, 36, and 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
percent
  Baseline | 8.6 (1.1) | 8.5 (1.9)
  Day 28: number analyzed (Participants) | 21 | 21
  Day 28 | 6.0 (0.6) | 6.1 (0.6)
  Day 84: number analyzed (Participants) | 21 | 17
  Day 84 | 4.8 (0.7) | 4.9 (0.3)
  Week 28: number analyzed (Participants) | 18 | 16
  Week 28 | 5.3 (1.3) | 5.2 (0.5)
  Week 36: number analyzed (Participants) | 18 | 17
  Week 36 | 5.3 (1.3) | 5.1 (0.6)
  Week 52: number analyzed (Participants) | 18 | 16
  Week 52 | 5.5 (1.6) | 5.3 (0.5)

13. Secondary Outcome: Fasting Blood Sugar (FBS) From Baseline (Pre-Transplant) Through Wk 52 Post-Transplant
Description: Fasting blood sugar (e.g., glucose) test is used to help diagnose diabetes, prediabetes, and gestational diabetes.
  Reference fasting blood sugar (glucose) values:
  * 70 to 99 mg/dL is normal
  * 100 to 125 mg/dL is considered prediabetes
  * 126 mg/dL or higher on two separate tests is considered diabetes.
Time Frame: Baseline (Pre-Transplant) and Days 28, 84, and Weeks 28, 36, and 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Investigational | Control
Number analyzed (Participants) | 21 | 19
mg/dL
  Baseline | 183.3 (107.2) | 217.3 (125.4)
  Day 28: number analyzed (Participants) | 21 | 18
  Day 28 | 100.0 (15.3) | 100.9 (20.5)
  Day 84: number analyzed (Participants) | 20 | 19
  Day 84 | 96.0 (44.9) | 89.7 (8.2)
  Week 28: number analyzed (Participants) | 21 | 18
  Week 28 | 106.5 (84.7) | 96.2 (22.6)
  Week 36: number analyzed (Participants) | 21 | 17
  Week 36 | 96.0 (27.8) | 87.2 (10.8)
  Week 52: number analyzed (Participants) | 20 | 19
  Week 52 | 98.6 (37.5) | 91.5 (12.1)

14. Secondary Outcome: Standardized Blood Pressure Measurement From Baseline (Pre-Transplant) Through Wk 52 Post-Transplant
Description: A blood pressure measurement consists of two numbers: the systolic and diastolic pressures. Systolic pressure measures the pressure in blood vessels when the heart beats. Diastolic pressure measures the pressure in blood vessels between beats of the heart.
  * Systolic measures of <120 and diastolic measures of <80 are considered normal.
  * Systolic measures of 120-139 and diastolic measures of 80-89 are considered at risk (or pre-hypertension).
  * Systolic measures of ≥140 and diastolic measures of ≥90 are considered high.
Time Frame: Baseline (Pre-Transplant) and Days 28, 84, and Weeks 28, 36, and 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
mmHg
  Systolic BP at Baseline | 161.3 (26.1) | 158.3 (23.7)
  Systolic BP at Day 28 | 116.9 (15.4) | 112.0 (16.8)
  Systolic BP at Day 84: number analyzed (Participants) | 22 | 19
  Systolic BP at Day 84 | 126.3 (19.2) | 123.8 (18.6)
  Systolic BP at Week 28: number analyzed (Participants) | 20 | 18
  Systolic BP at Week 28 | 136.1 (22.7) | 126.2 (23.8)
  Systolic BP at Week 36: number analyzed (Participants) | 19 | 19
  Systolic BP at Week 36 | 133.5 (20.5) | 126.7 (10.6)
  Systolic BP at Week 52: number analyzed (Participants) | 17 | 21
  Systolic BP at Week 52 | 132.0 (18.8) | 127.0 (15.4)
  Diastolic BP at Baseline | 82.7 (14.0) | 85.2 (10.5)
  Diastolic BP at Day 28 | 67.0 (8.4) | 65.4 (9.2)
  Diastolic BP at Day 84: number analyzed (Participants) | 22 | 19
  Diastolic BP at Day 84 | 72.8 (7.9) | 73.4 (10.1)
  Diastolic BP at Week 28: number analyzed (Participants) | 20 | 18
  Diastolic BP at Week 28 | 76.6 (8.8) | 73.3 (10.4)
  Diastolic BP at Week 36: number analyzed (Participants) | 19 | 19
  Diastolic BP at Week 36 | 76.5 (10.0) | 76.8 (8.8)
  Diastolic BP at Week 52: number analyzed (Participants) | 17 | 21
  Diastolic BP at Week 52 | 74.2 (8.6) | 77.0 (7.6)

15. Secondary Outcome: Count of Participants With Use of Anti-hypertensive Medication From Baseline (Pre-Transplant) Through Wk 52 Post-Transplant
Description: Anti-hypertensive medications are a class of drugs that are used to treat hypertension. The medications seek to prevent the complications of high blood pressure, such as stoke and myocardial infarction.
Time Frame: Baseline (Pre-Transplant) and Days 28, 84, and Weeks 28, 36, and 52
Population: Intent-to-treat population with available data
Measure: Number; unit: Count of Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Count of Participants
  Baseline | 18 | 19
  Day 28 | 14 | 10
  Day 84 | 11 | 7
  Week 28 | 13 | 11
  Week 36 | 13 | 11
  Week 52 | 13 | 11

16. Secondary Outcome: Fasting Lipid Profile at Baseline (Pre-Transplant)
Description: A fasting lipid profiles measures total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels. These measurements are used in assessing one's risk of cardiovascular disease. Target ranges for each of these measures are provided:
  * Total cholesterol: 75-169 mg/dL if age ≤20; 100-199 mg/dL if age ≥ 21; high values indicate risk of cardiovascular disease
  * LDL cholesterol: <70 mg/dL for people with documented cardiovascular disease or metabolic syndrome; <100 mg/dL for people considered high risk for cardiovascular disease; <130 mg/dL for people considered low risk for cardiovascular disease; high values indicate risk of cardiovascular disease
  * HDL cholesterol: 40mg/dL and higher; high values indicate reduced risk of cardiovascular disease
  * Non-HDL cholesterol: 30 mg/dL above the target value for LDL cholesterol; high values indicate risk of cardiovascular disease and
  * Triglycerides: <150 mg/dL; high values indicate risk of cardiovascular disease.
Time Frame: Baseline (Pre-Transplant)
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Investigational | Control
Number analyzed (Participants) | 19 | 19
mg/dL
  Tot. Chol. Baseline | 142.8 (38.1) | 140.5 (42.0)
  Non-HDL Baseline | 91.0 (28.0) | 82.4 (42.0)
  LDL Baseline | 66.5 (28.0) | 60.7 (32.9)
  HDL Baseline | 51.8 (19.0) | 58.1 (16.2)
  Triglyc. Baseline | 120.9 (55.2) | 107.5 (55.1)

17. Secondary Outcome: Fasting Lipid Profile at Wk 28 Post-Transplant
Description: as for outcome 16
Time Frame: Week 28 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Investigational | Control
Number analyzed (Participants) | 17 | 16
mg/dL
  Tot. Chol. Week 28 | 159.9 (48.8) | 149.2 (28.7)
  Non-HDL Week 28 | 112.6 (45.4) | 97.4 (27.9)
  LDL Week 28 | 93.1 (43.9) | 81.2 (28.5)
  HDL Week 28 | 47.3 (15.1) | 51.8 (11.8)
  Triglyc. Week 28 | 93.2 (52.6) | 87.8 (44.1)

18. Secondary Outcome: Lipid Profile at Wk 52 Post-Transplant
Description: A fasting lipid profiles measures total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels. These measurements are used in assessing one's risk of cardiovascular disease. Target ranges for each of these measures are provided:
  * Total cholesterol: 75-169 mg/dL if age ≤ 20; 100-199 mg/dL if age ≥ 21; high values indicate risk of cardiovascular disease
  * LDL cholesterol: <70 mg/dL for people with documented cardiovascular disease or metabolic syndrome; <100 mg/dL for people considered high risk for cardiovascular disease; <130 mg/dL for people considered low risk for cardiovascular disease; high values indicate risk of cardiovascular disease
  * HDL cholesterol: 40mg/dL and higher; high values indicate reduced risk of cardiovascular disease
  * Non-HDL cholesterol: 30 mg/dL above the target value for LDL cholesterol; high values indicate risk of cardiovascular disease and
  * Triglycerides: <150 mg/dL; high values indicate risk of cardiovascular disease.
Time Frame: Week 52 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Investigational | Control
Number analyzed (Participants) | 19 | 13
mg/dL
  Tot. Chol. Week 52 | 164.2 (38.9) | 162.8 (44.1)
  Non-HDL Week 52: number analyzed (Participants) | 19 | 12
  Non-HDL Week 52 | 115.7 (38.1) | 112.3 (38.5)
  LDL Week 52: number analyzed (Participants) | 19 | 12
  LDL Week 52 | 96.9 (36.5) | 92.7 (33.1)
  HDL Week 52: number analyzed (Participants) | 19 | 12
  HDL Week 52 | 48.5 (16.7) | 47.3 (12.8)
  Triglyc. Week 52: number analyzed (Participants) | 19 | 12
  Triglyc. Week 52 | 88.6 (34.9) | 95.4 (75.0)

19. Secondary Outcome: Count of Participants With Use of Lipid Lowering Medications at Baseline, Wk 28 and Wk 52 Post-Transplant
Description: Lipid lowering medications are used in the treatment of high levels of fats (lipids), such as cholesterol in blood
Time Frame: Baseline (Pre-Transplant), Week 28, and Week 52
Population: Intent-to-treat population
Measure: Number; unit: participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
participants
  Baseline | 18 | 18
  Week 28 | 19 | 16
  Week 52 | 19 | 16

20. Secondary Outcome: Count of Participants With Acute Rejection (AR) of Kidney or Pancreatic Transplant During the First 52 Wks Post-Transplant
Description: Biopsy-proven acute rejection (AR) of the kidney (renal) or pancreas during the first 52 weeks post-transplant. AR grading using standard Banff* criteria. For both kidney and pancreas, AR is defined as a grade ≥1.
  * AR for the kidney: Banff 2007 criteria. Severity of AR is graded by as IA, IB, IIA, IIB, or III, with IA defined as the mildest form of AR and III being the most severe.
  * AR for the pancreas: Banff 2011 Criteria. Severity of AR is graded as I, II, or III, with I defined as the mildest form of AR and III being the most severe.
Time Frame: Transplant through Week 52
Population: Intent-to-treat population
Measure: Number; unit: Count of Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Count of Participants
  Kidney | 2 | 2
  Pancreas | 5 | 1

21. Secondary Outcome: Severity Grade of First Biopsy-Proven Acute Rejection (AR) During the First 52 Weeks Post-Transplant
Description: AR grading using standard Banff* criteria. For both kidney and pancreas, AR is defined as a grade ≥1.
  * AR for the kidney: Banff 2007 criteria. Severity of AR is graded by as IA, IB, IIA, IIB, or III, with IA defined as the mildest form of AR and III being the most severe.
  * AR for the pancreas: Banff 2011 Criteria. Severity of AR is graded is I, II, or III, with I defined as the mildest form of AR and III being the most severe.
Time Frame: Transplant through Week 52
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants
  Kidney First Grade IA | 0 | 1
  Kidney First Grade IB | 1 | 0
  Kidney First Grade IIA | 0 | 1
  Kidney First Grade IIB | 1 | 0
  Pancreas First Grade I | 4 | 0
  Pancreas First Grade II | 1 | 1

22. Secondary Outcome: Count of Participants With Biopsy-Proven Humoral Rejection During the First 52 Weeks Post-Transplant
Description: Humoral rejection (i.e., antibody mediated rejection) of:
  1. the kidney as defined by diffusely positive staining for C4d, presence of circulating anti-donor antibodies, and morphologic evidence of acute tissue injury determined by local pathology and,
  2. the pancreas as defined by the presence of circulating anti-donor antibodies, and histopathological data including morphologic evidence of microvascular tissue injury and C4d staining in interacinar capillaries determined by local pathology.
Time Frame: Transplant through Week 52
Population: Intent-to-treat population with available data
Measure: Number; unit: Count of Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Count of Participants
  Kidney | 0 | 0
  Pancreas | 0 | 0

23. Secondary Outcome: Count of Participants With De Novo Anti-Donor Antibodies or Anti-Human Leukocyte Antigen (HLA) Antibodies During the First 52 Weeks Post-Transplant
Description: The de novo development of donor-specific antibody (DSA) is associated with an increased risk of graft rejection.
  The presence of anti-Histocompatibility Antigen (HLA) antibodies (alloantibodies) is associated with increased risk of acute and chronic injury to the transplant allograft.
Time Frame: Transplant through Week 52
Population: Intent-to-treat population with available data
Measure: Number; unit: Count of Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 20
Count of Participants
  De novo DSA | 0 | 0
  Anti-HLA | 2 | 1

24. Secondary Outcome: Type of Treatment(s) Participants Received for Biopsy-Proven Renal Allograft Rejection During the First 52 Weeks Post-Transplant
Description: Participants are stratified by kidney biopsy results/treatment received.
  In the event of a for cause renal (kidney) biopsy:
  -The diagnosis of acute cellular rejection (ACR) using the Banff 2007 renal allograft pathology criteria. These criteria for renal allograft biopsies is an international histopathological classification standard. ACR is defined by a renal biopsy demonstrating a Banff 2007 classification of Grade IA or greater, with higher scores indicating more severe rejection. (Ref: Solez K, Colvin RB et al. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant 2008 8(4): 753-60).
  Acronyms and abbreviations:
  * ACR=Acute Cellular Rejection*
  * Normal*
  * Borderline* (criteria for ACR not fulfilled)
  * Gd.=Grade*
  * IFTA=Interstitial Fibrosis and Tubular Atrophy*
  * ATG=Anti-thymocyte globulin therapy
  * IVIG=Intravenous Immunoglobulin therapy
  * PO=Orally
  * QD=Daily *Banff 2007 renal allograft pathology criteria
Time Frame: Transplant through Week 52
Population: Intent-to-treat population with available data. All participants were considered evaluable for rejection. Only 'for cause' biopsies were performed post-transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants
  Borderline/None: number analyzed (Participants) | 11 | 11
  Borderline/None | 1 | 0
  Borderline/Pulse Steroids: number analyzed (Participants) | 11 | 11
  Borderline/Pulse Steroids | 0 | 1
  Borderline, IFTA-Gd. I/Pulse Steroids, IVIG: number analyzed (Participants) | 11 | 11
  Borderline, IFTA-Gd. I/Pulse Steroids, IVIG | 0 | 1
  ACR-Gd. IA/ATG, Pulse Steroids: number analyzed (Participants) | 11 | 11
  ACR-Gd. IA/ATG, Pulse Steroids | 0 | 1
  ACR-Gd. IB/ATG, Pulse Steroids: number analyzed (Participants) | 11 | 11
  ACR-Gd. IB/ATG, Pulse Steroids | 1 | 0
  ACR-Gd. IIA/ATG, Pulse Steroids: number analyzed (Participants) | 11 | 11
  ACR-Gd. IIA/ATG, Pulse Steroids | 0 | 1
  ACR-Gd. IIB/ATG, Pulse Steroids: number analyzed (Participants) | 11 | 11
  ACR-Gd. IIB/ATG, Pulse Steroids | 1 | 0
  IFTA-Gd. I/None: number analyzed (Participants) | 11 | 11
  IFTA-Gd. I/None | 1 | 0
  IFTA-Gd. I/Potassium citrate: number analyzed (Participants) | 11 | 11
  IFTA-Gd. I/Potassium citrate | 2 | 0
  Normal/Steroids QD: number analyzed (Participants) | 11 | 11
  Normal/Steroids QD | 0 | 1
  No grade reported/IVIG: number analyzed (Participants) | 11 | 11
  No grade reported/IVIG | 1 | 0
  No grade reported/None | 1 | 4
  Normal/None | 3 | 2

25. Secondary Outcome: Type of Treatment(s) Participants Received for Biopsy-Proven Pancreatic Allograft Rejection During the First 52 Weeks Post-Transplant
Description: Participants are stratified by kidney biopsy results/treatment received.
  Upon having a for-cause biopsy performed, persons often receive treatment for rejection based on the biopsy results, which may or may not reveal signs of rejection. Details of biopsy findings and corresponding treatment are provided for each instance of treatment for rejection.
  Results summary format: biopsy results; treatment.
  Acronyms and abbreviations:
  * ACR=Acute Cellular Rejection
  * IFTA=Interstitial Fibrosis and Tubular Atrophy
  * ATG=Anti-thymocyte globulin therapy
  * IVIG=Intravenous Immunoglobulin therapy
  * Gd =Grade
  * PO=Orally
  * QD=Daily
Time Frame: Transplant through Week 52
Population: Intent-to-treat population with available data. Only 'for cause' biopsies were performed post-transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants
  ACR-Gd. I/ATG: number analyzed (Participants) | 6 | 1
  ACR-Gd. I/ATG | 1 | 0
  ACR-Gd. I/ATG, Pulse Steroids: number analyzed (Participants) | 6 | 1
  ACR-Gd. I/ATG, Pulse Steroids | 1 | 0
  ACR-Gd. I/ATG, Pulse Steroids, IVIG: number analyzed (Participants) | 6 | 1
  ACR-Gd. I/ATG, Pulse Steroids, IVIG | 1 | 0
  ACR-Gd. I, IFTA-Gd. I/Pulse Steroids, Solumedrol,: number analyzed (Participants) | 6 | 1
  ACR-Gd. I, IFTA-Gd. I/Pulse Steroids, Solumedrol, | 1 | 0
  ACR-Gd. II/ATG, Pulse Steroids: number analyzed (Participants) | 6 | 1
  ACR-Gd. II/ATG, Pulse Steroids | 1 | 1
  No grade reported/None | 1 | 0

26. Secondary Outcome: Count of Participants With Event of Death, Graft Loss, or Undetectable C-peptide
Description: This measure counts death, graft loss, or undetectable C-peptide value (e.g., C-peptide <0.3 ng/mL) occurring at any point post-transplant and independent of each other.
  * Kidney Graft Loss was defined as 90 consecutive days of dialysis dependency.
  * Pancreas graft loss was defined as returning to exogenous insulin therapy or initiation of oral hypoglycemic agents for greater than 30 days.
  * Factitious hypoglycemia due to surreptitious insulin administration results in elevated serum insulin levels and low or undetectable C-peptide levels.
Time Frame: Transplant through Week 52 Post-Transplant
Population: Intent-to-treat population with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants
  Death | 1 | 0
  Kidney Graft Loss | 0 | 0
  Pancreas Graft Loss | 1 | 0
  Undetectable C-peptide | 0 | 0

27. Secondary Outcome: Count of Participants With the Occurrence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse events were collected systematically. Counts of all participants who experienced at least one adverse event (AEs, SAEs) by assigned treatment group.
  Refer to the Serious Adverse Events and Other Adverse Events tables for more detail.
Time Frame: From Enrollment (Pre-Transplant) to Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Number; unit: Count of Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Count of Participants
  All Adverse Events | 22 | 21
  Serious Adverse Events | 20 | 19

28. Secondary Outcome: Count of Participants With an Infectious Disease Serious Adverse Event(s) Requiring Hospitalization or Systemic Therapy
Description: Infections were required to be reported as a serious adverse event if they required either inpatient hospitalization or prolongation of a current hospitalization. Displayed are counts of all participants who experienced infection(s) as an adverse event, by treatment group.
Time Frame: Transplant through Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants | 11 | 11

29. Secondary Outcome: Count of Participant Diagnosed With BK Polyoma Virus (BKV) and Cytomegalovirus (CMV) Viremia As Adverse Events
Description: Viral infections following renal transplantation is a significant source of recipient morbidity and mortality, and a significant cause of allograft dysfunction and loss.
  Specific viruses were monitored during this study using participant blood samples. Displayed are counts of participants who experienced BKV and CMV viremia as adverse events, diagnosed by test results from the local clinical pathology laboratory.
Time Frame: Transplant through Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Number; unit: Count of Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Count of Participants
  BK Viremia | 8 | 3
  CMV Viremia | 5 | 3

30. Secondary Outcome: Count of Participants Diagnosed With Epstein-Barr Virus (EBV) Infection as an Adverse Event
Description: Viral infections following renal transplantation is a significant source of recipient morbidity and mortality, and a significant cause of allograft dysfunction and loss. Specific viruses were monitored during this study using participant blood samples. Displayed are counts of all participants diagnosed with EBV infection as an adverse event by EBV test(s), diagnosed by test results from the local clinical pathology laboratory.
Time Frame: Transplant through Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

31. Secondary Outcome: Count of Participants Diagnosed With Malignancy as an Adverse Event
Description: An increased risk/incidence of malignancy is a recognized complication of immunosuppression in recipients of organ transplants. In Phase 3 clinical trials, overall malignancy rates were similar across all treatment groups, with the exception of posttransplant lymphoproliferative disease (PTLD).Displayed are counts of all participants who experienced malignancy reported as an adverse event.
Time Frame: Transplant through Week 52 Post-Transplant
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Transplantation until end of study (up to 76 weeks)
Arm/Group | Investigational | Control | Enrolled, Not Randomized
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/21 | 0/3
Serious Adverse Events (participants affected / at risk) | 20/22 | 19/21 | 0/3
Other Adverse Events (participants affected / at risk) | 20/22 | 19/21 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=22) | Control (N=21) | Enrolled, Not Randomized (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Pancreas transplant rejection (Immune system disorders) | 7 (7) | 3 (4) | 0 (0)
Renal and pancreas transplant rejection (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancreatic abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (6) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Renal transplant torsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=22) | Control (N=21) | Enrolled, Not Randomized (N=3)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 10 (11) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 6 (7) | 3 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
BK virus infection (Infections and infestations) | 8 (8) | 3 (3) | 0 (0)
Clostridial infection (Infections and infestations) | 2 (2) | 3 (4) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 3 (6) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (12) | 3 (4) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 3 (4) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT01790594/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT01790594/ICF_001.pdf